CLINICAL TRIAL: NCT05142696
Title: A Phase Ib/II Dose Finding Study Assessing Safety and Efficacy of [177Lu]Lu-DOTA-TATE in Newly Diagnosed Extensive Stage Small Cell Lung Cancer (ES-SCLC) in Combination With Carboplatin, Etoposide, and Atezolizumab in Induction and With Atezolizumab in Maintenance Phase
Brief Title: A Study of [177Lu]Lu-DOTA-TATE in Newly Diagnosed ES-SCLC Patients in Combination With Carboplatin, Etoposide and Atezolizumab
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAAA601A42101; 2021-004155-16 (EudraCT Number); 2024-513185-19-00 (Other: EU CTIS)
Record Dates: First submitted 2021-11-15; First posted 2021-12-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: Extensive Stage Small Cell Lung Cancer; ES-SCLC; Radioligand therapy; RLT; [177Lu]Lu-DOTA-TATE; Lutathera; Lutetium (177Lu) oxodotreotide; Lutetium Lu 177 dotatate; atezolizumab; carboplatin; etoposide
MeSH Terms: interventions — lutetium Lu 177 dotatate; atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Level 1 (DL1) (Experimental): Dose Level 1 (DL1): [177Lu]Lu-DOTA-TATE 100 mCi with carboplatin AUC 5 D1, etoposide 100 mg/m2 D1-3, and atezolizumab 1200 mg in induction period, then [177Lu]Lu-DOTA-TATE 100 mCi plus atezolizumab 1200 mg in the maintenance period.
  Interventions: Drug: [177Lu]Lu-DOTA-TATE; Drug: Atezolizumab; Drug: [68Ga]Ga-DOTA-TATE; Other: Carboplatin; Other: Etoposide
- Dose Level 2a (DL2a) (Experimental): Dose Level 2a (DL2a): [177Lu]Lu-DOTA-TATE 150 mCi with carboplatin AUC 5 D1, etoposide 100 mg/m2 D1-3 and atezolizumab 1200 mg in induction period, then [177Lu]Lu-DOTA-TATE 150 mCi plus atezolizumab 1200 mg in the maintenance period.
  Interventions: Drug: [177Lu]Lu-DOTA-TATE; Drug: Atezolizumab; Drug: [68Ga]Ga-DOTA-TATE; Other: Carboplatin; Other: Etoposide
- Dose Level 2b (DL2b) (Experimental): Dose Level 2b (DL2b): [177Lu]Lu-DOTA-TATE 150 mCi with carboplatin AUC 5 D1, etoposide 100 mg/m2 D1-3 and atezolizumad 1200 mg in induction period, then [177Lu]Lu-DOTA-TATE 200 mCi plus atezolizumab 1200 in the maintenance period.
  Interventions: Drug: [177Lu]Lu-DOTA-TATE; Drug: Atezolizumab; Drug: [68Ga]Ga-DOTA-TATE; Other: Carboplatin; Other: Etoposide
- Dose Level 3a (DL3a) (Experimental): Dose Level 3a (DL3a): [177Lu]Lu-DOTA-TATE 200 mCi with carboplatin AUC 5 D1, etoposide 100 mg/m2 D1-3, and atezolizumab 1200 mg in induction period, then [177Lu]Lu-DOTA-TATE 200 mCi plus atezolizumab 1200 mg in the maintenance period.
  Interventions: Drug: [177Lu]Lu-DOTA-TATE; Drug: Atezolizumab; Drug: [68Ga]Ga-DOTA-TATE; Other: Carboplatin; Other: Etoposide
- Dose Level 3b (DL3b) (Experimental): Dose Level 3b (DL3b): [177Lu]Lu-DOTA-TATE 200 mCi with carboplatin AUC 5 D1, etoposide 100 mg/m2 D1-3, and atezolizumab 1200 mg in induction period, then [177Lu]Lu-DOTA-TATE 250 mCi plus atezolizumab 1200 mg in the maintenance period.
  Interventions: Drug: [177Lu]Lu-DOTA-TATE; Drug: Atezolizumab; Drug: [68Ga]Ga-DOTA-TATE; Other: Carboplatin; Other: Etoposide
- Dose Level 4 (DL4) (Experimental): Dose Level 4 (DL4): [177Lu]Lu-DOTA-TATE 250 mCi with carboplatin AUC 5 D1, etoposide 100 mg/m2 D1-3 and atezolizumab 1200 mg in induction period, then [177Lu]Lu-DOTA-TATE 250 mCi plus atezolizumab 1200 mg in the maintenance period.
  Interventions: Drug: [177Lu]Lu-DOTA-TATE; Drug: Atezolizumab; Drug: [68Ga]Ga-DOTA-TATE; Other: Carboplatin; Other: Etoposide
- Phase II Experimental arm (Experimental): [177Lu]Lu-DOTA-TATE at recommended dose declared in phase I part in combination with carboplatin, etoposide and atezolizumab (experimental arm)
  Interventions: Drug: Atezolizumab; Drug: [68Ga]Ga-DOTA-TATE; Other: Carboplatin; Other: Etoposide
- Phase II Control arm (Other): Carboplatin, etoposide and atezolizumab alone (control arm)
  Interventions: Drug: Atezolizumab; Drug: [68Ga]Ga-DOTA-TATE; Other: Carboplatin; Other: Etoposide

INTERVENTIONS:
Drug: [177Lu]Lu-DOTA-TATE — Solution for infusion of [177Lu]Lu-DOTA-TATE will be administered as follows:
  * 2 administrations during the induction period on either Day 3, 4 or 5 of Week 1 and on Week 7 Day 3
  * 1 to 4 administrations during the maintenance period on Week 13 Day 1, Week 16 Day 1, Week 19 Day 1 and Week 22 Day 1, depending on the dose assessed
  Other Names: Lutathera; Lutetium (177Lu) oxodotreotide; Lutetium Lu 177 dotatate
  Arms: Dose Level 1 (DL1); Dose Level 2a (DL2a); Dose Level 2b (DL2b); Dose Level 3a (DL3a); Dose Level 3b (DL3b); Dose Level 4 (DL4)
Drug: Atezolizumab — Atezolizumab 1200 mg on Day 1 from Cycle 2 every 3 weeks in induction and maintenance period
Drug: [68Ga]Ga-DOTA-TATE — 2 MBq/kg of body weight (0.054 mCi/kg), with a minimum dose of 100 MBq (2.7 mCi) and maximum dose of 200 MBq (5.4 mCi)
Other: Carboplatin — Four cycles of carboplatin AUC 5 on Day 1 every 3 weeks (Weeks 1, 4, 7 and 10) in induction period
Other: Etoposide — Four cycles of etoposide 100 mg/m2 on Day 1-3, every 3 weeks (Weeks 1, 4, 7 and 10) in induction period

SUMMARY:
This study aims to establish a safe and well tolerated dose of [177Lu]Lu-DOTA-TATE in combination with carboplatin, etoposide and atezolizumab in this setting and to assess preliminary efficacy of this combination treatment versus the combination of carboplatin, etoposide, and atezolizumab.The study will be essential to assess a new potential therapeutic option in participants with this aggressive cancer type.

DETAILED DESCRIPTION:
The study for each participant consists of a Screening period, a Treatment period that includes an Induction treatment period and a Maintenance treatment period, and a Follow-up period.

The study will consist of a Phase Ib dose escalation with concurrent backfill part and a randomised controlled Phase II part.

During the screening period of up to 28 days before starting SCLC treatment, each participant will be assessed for somatostatin receptor (SSTR) expression by [68Ga]Ga-DOTA-TATE imaging PET/scan.

The dose escalation part in this study will be guided by the dose limiting toxicity (DLT) rate observed during the DLT period. To achieve a more robust dataset and to aid dose decisions, additional participants may be backfilled in each dose level.

Upon declaring RD, a 1:1 randomised Phase II with approximately 140 participants with newly diagnosed ES-SCLC will be enrolled and receive either [177Lu]Lu-DOTA-TATE at the RD in combination with carboplatin, etoposide and atezolizumab (experimental arm) or carboplatin, etoposide and atezolizumab alone (control arm).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is >= 18 years on the day of signing informed consent form
* Histologically or cytologically confirmed ES-SCLC
* Presence of measurable disease
* No prior systemic treatment for ES-SCLC (except the first cycle of chemotherapy with or without atezolizumab of the induction period
* ECOG status =< 1
* Provision of tumor tissue to support exploratory biomarker analysis
* Life expectancy of >= 6 months

Key Exclusion Criteria:

* Participant has received prior therapy with an antibody or drug against immune checkpoint pathways
* Active autoimmune diseases or history of autoimmune diseases that may relapse
* Severe chronic or active infections (including active tuberculosis, HBV, or HCV infection) requiring systemic antibacterial, antifungal or antiviral therapy within 2 weeks before Cycle 1 Day 1
* Any major surgical procedure requiring general anesthesia =< 28 days before Cycle 1 Day 1
* History or current diagnosis of electrocardiogram (ECG) abnormalities indicating significant risk of safety for participants participating in the study
* Known hypersensitivity to the active substances or any of the excipients of the study drugs
* Concurrent participation in another therapeutic clinical study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2029-03-09 (Estimated); Study Completion 2029-03-23 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Frequency of dose limiting toxicities (DLTs), Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs leading to treatment discontinuation | Within the first six weeks of [177Lu]Lu-DOTA-TATE treatment]
  A dose-limiting toxicity (DLT) is defined as an AE or abnormal laboratory value assessed as unrelated to disease, disease progression, intercurrent illness, or concomitant medications with an onset within the first cycle of initiation of [177Lu]Lu-DOTA-TATE treatment. The National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) version 5.0 will be used for AE grading.
Phase ll: Overall survival (OS) | In the phase II part: From date of randomization until date of death from any cause, assessed up to 3 years (estimated final Overall Survival (OS) analysis)
  To assess efficacy of [177Lu]Lu-DOTA-TATE in combination with atezolizumab, carboplatin, and etoposide (experimental arm) versus standard of care consisting of carboplatin, etoposide, and atezolizumab (control arm) in terms of overall survival

SECONDARY OUTCOMES:
Phase lb: Objective Response Rate (ORR) based on Investigator assessment | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed for up to 3 years (estimated final Overall Survival (OS) analysis)
  Objective Response Rate (ORR) defined as the proportion of participants with a best overall confirmed complete response (CR) or partial response (PR) as assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by Investigator assessment
Phase lb: Duration of Response (DOR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed for up to 3 years (estimated final Overall Survival (OS) analysis)
  Duration of Response (DOR), calculated as the time from the date of the first documented CR or PR to the first documented progression or death due to underlying cancer. Participants continuing without progression or death due to underlying cancer will be censored at the date of their last adequate tumor assessment. DOR will be listed and summarized by dose level combination and checkpoint inhibitor in Phase Ib and by treatment group in Phase II part for all participants in the FAS with confirmed BOR of CR or PR.
Phase lb: Progression Free Survival (PFS) based on Investigator assessment | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed for up to 3 years (estimated final OS analysis)
  Progression Free Survival (PFS) is defined as the time from the date of first dose to the date of the first documented progression or death due to any cause. PFS will be assessed via local review according to RECIST 1.1. If no PFS event is observed, PFS will be censored at the date of the late adequate tumor assessment prior to data cut-off date and start of new anti-neoplastic therapy, whichever comes first.
  PFS will be analyzed in the FAS population according to the assigned dose level combination and checkpoint inhibitor in Phase Ib and by treatment group in Phase II part. The PFS distribution will be estimated using the Kaplan-Meier method, and the Kaplan-Meier curves, medians and 95% confidence intervals of the medians will be presented for each dose level combination and checkpoint inhibitor in Phase Ib and by treatment group in Phase II part.
Phase lb: Overall Survival (OS) | From date of randomization until date of death from any cause, assessed up to 3 years (estimated final Overall Survival (OS) analysis)
  OS is defined as the time from date of first dose to date of death due to any cause in Phase Ib. If a participant is not known to have died, then OS will be censored at the latest date the participant was known to be alive (on or before the cut-off date).
  OS will be analyzed in the FAS population according to the assigned dose cohort and checkpoint inhibitor in Phase Ib. The OS distribution will be estimated using the Kaplan-Meier method, and the Kaplan-Meier curves, medians and 95% confidence intervals of the medians will be presented for each dose level combination and checkpoint inhibitor in Phase Ib Kaplan-Meier estimates with 95% confidence intervals every 6 months will be summarized as well by dose level combination, checkpoint inhibitor in Phase Ib and treatment group in Phase II part.
Phase ll: Progression free survival (PFS) by investigator assessment | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed for up to 3 years (estimated final OS analysis)
  Progression Free Survival (PFS) is defined as the time from the date of first dose to the date of the first documented progression or death due to any cause. PFS will be assessed via local review according to RECIST 1.1. If no PFS event is observed, PFS will be censored at the date of the late adequate tumor assessment prior to data cut-off date and start of new anti-neoplastic therapy, whichever comes first.
Phase ll: Objective Response Rate (ORR) by investigator assessment | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed for up to 3 years (estimated final Overall Survival (OS) analysis)
  Objective response rate (ORR) is defined as the percentage of participants with confirmed best overall confirmed complete response (CR) or partial response (PR), as per local review and according to RECIST 1.1 by Investigator assessment.
Phase ll: Duration of Response (DOR) by investigator assessment | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed for up to 3 years (estimated final Overall Survival (OS) analysis)
  Duration of Response (DOR), calculated as the time from the date of the first documented CR or PR to the first documented progression or death due to underlying cancer. Participants continuing without progression or death due to underlying cancer will be censored at the date of their last adequate tumor assessment. DOR will be listed and summarized by dose level combination and checkpoint inhibitor in Phase Ib and by treatment group in Phase II part for all participants in the FAS with confirmed BOR of CR or PR.
Incidence and severity of adverse events (AEs), serious AEs (SAEs), changes in hematology and chemistry values, vital signs, and ECGs; dose interruptions, discontinuations, and reductions | From date of randomisation until date of progression or date of death from any cause, whichever comes first, assessed for up to 3 years
  To characterize the safety and tolerability of [177Lu]Lu-DOTA-TATE in combination with carboplatin, etoposide, and atezolizumab in induction treatment and with atezolizumab in maintenance treatment in newly diagnosed participants with ES-SCLC
Incidence and severity of Adverse Events (AEs) and serious Adverse Events (SAEs) within 48 hours after [68Ga]Ga-DOTA-TATE infusion | up to 48 hours following the start of [68Ga]Ga-DOTA-TATE administration]
  To assess the safety and tolerability of [68Ga]Ga-DOTA-TATE in participants with newly diagnosed ES-SCLC
Phase lb and II: Absorbed radiation doses of [177Lu]Lu-DOTA-TATE | Week 7 Day 3
  To characterize the pharmacokinetics (PK) and dosimetry of [177Lu]Lu-DOTA-TATE in participants with newly diagnosed ES-SCLC
Phase lb: PK parameters of [177Lu]Lu-DOTA-TATE in blood | Week 7 Day 3 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 7 Day 4 (24 hours post-dose), Week 7 Day 5 (48 hours post-dose), Week 8 Day 3 (168 hours post-dose)
  Blood samples for radioactivity measurement will be collected in all participants who undergo dosimetry assessments (i.e. first 3 participants at dose levels 1, 2a or 2b, 3a or 3b, and 4). For the rest of participants , blood samples will be taken before the start of [177Lu]Lu-DOTA-TATE infusion, at the end of infusion, and then at 2h, 6h after the end of [177Lu]Lu-DOTA-TATE infusion. Blood samples will be drawn in heparinized tubes. Radioactivity measurements on blood will be performed locally on site, using a gamma-counter.
Phase II: PK parameters of [177Lu]Lu-DOTA-TATE in blood | Week 1 Day 3, Week 7 Day 3 (pre-dose, before the end of infusion, post-dose: 2 hours, 6 hours, 24 hours, 48 hours, 168 hours), Week 13 Day 1 (pre-dose, before the end of infusion, post-dose: 2 hours, 6 hours, 24 hours, 48 hours post-dose)
  Blood samples for radioactivity measurement will be collected in approximately 10 participants who undergo dosimetry assesments. In the participants that will undergo dosimetry assessments, an additional whole body planar transmission scan with the participant needs to be performed for the qualification of the dosimetry setup before the first infusion of [177Lu]Lu-DOTA-TATE.
  A SPECT/CT scan will be acquired after the 1st, 2nd, and 4th administration of [177Lu]Lu-DOTA-TATE.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- United States (9):
  - Georgetown University Lombardi Cancer Center, Washington D.C., District of Columbia
  - Advent Health Cancer Institute, Orlando, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - University of Kentucky, Lexington, Kentucky
  - St. Louis University, St Louis, Missouri
  - Hackensack Meridian Health, Edison, New Jersey
  - University Hospitals Of Cleveland, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Ctr, Nashville, Tennessee
- Austria (3):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz, Upper Austria
  - Novartis Investigative Site, Vienna
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- China (2):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Olomouc, Czechia
- France (6):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Villejuif
- Germany (2):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Hong Kong, Hong Kong
- Israel (4):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Napoli
- Netherlands (2):
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (4):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
- Taiwan (3):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No